CLINICAL TRIAL: NCT03630068
Title: Stereotactic Image-Guided Microwave Ablation for Hepatocellular Carcinoma - Does Computer-assistance Broaden Eligibility and Efficacy of Ablative Treatment?
Brief Title: Computer-assisted Tumor Ablation for Patients With Liver Cancer
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SIGMAHCC_1
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Neoplasms; Hepatocellular Carcinoma; Ablation Techniques; Stereotaxic Techniques; Computer-Assisted Therapy; Computer-Assisted Surgery; Interventional Radiology
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hepatocellular carcinoma treated with microwave
  Interventions: Procedure: Stereotactic percutaneous image-guided microwave ablation

INTERVENTIONS:
Procedure: Stereotactic percutaneous image-guided microwave ablation — Stereotactic percutaneous image-guided microwave ablation implies the use of computer-assisted navigation technology for 3D trajectory planning and stereotactic placement of ablation probes, before applying local microwave ablation therapy

SUMMARY:
In patients with primary liver cancer arising from the liver cells, several treatment options are available according to the stage of the disease. Thermal ablation is a treatment modality using the deposition of thermal energy via an ablation probe to locally destroy the tumor tissue. It has been accepted as being equally effective as surgical resection in patients with very small tumors, as well as for patients with more advanced disease who are not surgical candidates or who are awaiting liver transplantation. Treatment success of thermal ablation is linked to the completeness of the tumor ablation and thus to the precision with which the ablation probes can be placed within the tumors. In recent years, novel computer-assister technology has been introduced to augment accuracy in ablation probe positioning, and first reports describing the safety and efficiency of these procedures have been described in the literature. However, very few works describe the oncological outcomes of patients when using this technology for thermal ablation. In this study, the investigators aim to describe local tumor control and the oncological follow-up of patients when using computer-assisted technology for thermal ablation of liver cancer.

DETAILED DESCRIPTION:
Curative treatment options for patients with early-stage hepatocellular carcinoma (HCC) include surgical resection, liver transplantation and local ablation. While only 20-25% of patients with HCC qualify for surgical resection or liver transplantation, local thermal ablation using radiofrequency or microwave energy represents a more tissue-sparing therapy with promising results. Thermal ablation has been accepted as valid alternative to resection in patients with very small solitary tumors (BCLC stage 0) with equally good survival rates up to 75 % at 5 years. It further represents a valid treatment modality for patients with limited tumor burden (BCLC stage A) who are not surgical candidates due to associated comorbidities. More recently, indications for thermal ablation have also been widened for patients with more advanced disease but still limited tumor burden (BCLC stage B1), as well as for use within combined treatment strategies and as bridging therapy in patients awaiting liver transplantation.

The major advantage of thermal ablation lies in its tissue-sparing yet locally destructive therapeutic character, which when combined with a minimally invasive access leads to low treatment-associated tissue trauma and morbidity. Regarding treatment efficiency, initial complete response is an independent predictive factor for survival for HCC patients treated with ablation. Hence, the precision of ablative therapy is crucial for treatment success, and relies directly on the accuracy of ablation probes positioning within the tumor target. To address this issue, advanced image-guided navigation technology has been introduced for use in liver-directed therapies. While first works reporting on the safety and accuracy of stereotactic percutaneous image-guided ablation of liver tumors are available, only few studies reporting on the oncological outcomes in liver tumors exist. No data on the oncological follow-up after stereotactic image-guided ablation of HCC is available to date, leaving the understanding of the clinical impact when using such novel navigation technology for ablative treatment in these patients scarce.

Overall, the investigators hypothesize that stereotactic image-guided microwave ablation allows a more precise and thus effective ablative treatment of HCC when compared to using conventional image-guidance techniques. This is due to the possibility of i) planning of targeting trajectories even for difficult-to-target lesions, ii) placement of ablation probes in multiple parallel needle configurations for larger lesions, iii) immediate intraoperative knowledge of treatment success through overlapping of pre- and post-ablation images with the possibility of re-ablation, and iv) reproducibility and standardization of the treatment technique. In this first retrospective analysis, the investigators aim to report therapeutic efficacy in terms local tumor control and short-term survival when using stereotactic image-guided microwave ablation for treatment of HCC, and further report procedural efficiency in terms of targeting accuracy and required time consumption.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent stereotactic percutaneous image-guided microwave ablation of hepatocellular carcinoma from 01.01.2015 to 31.12.2017 at Inselspital University Hospital of Bern Switzerland

Exclusion Criteria:

* Lack of general consent for data usage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma deemed amenable to percutaneous microwave ablation at the Multi-Disciplinary Team conference of the Department of Visceral Surgery and Medicine of the University Hospital of Bern, Switzerland
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | Through study completion, an average of 1 year
  Kaplan-Meier method
Recurrence-free survival | Through study completion, an average of 1 year
  Kaplan-Meyer method. Local recurrence defined as radiological suspicion of active tumor tissue within 10mm of the ablated lesions

SECONDARY OUTCOMES:
Local tumor progression rate | Through study completion, an average of 1 year
  Number of patients with local recurrences
Need for further liver-specific treatment | Through study completion, an average of 1 year
  Number and type of re-interventions (ablations, resections, transplantation)
Accuracy of ablation probe positioning | Intraoperative
  Deviation of ablation probe position as compared to planned ablation probe trajectory in the navigation system, reported in millimeters
Procedural efficiency | Intraoperative
  Time for planning/targeting/validation process of procedure and overall duration of procedure, reported in minutes
Clinical and radiological complications | At 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Tinguely, MD, Principal Investigator — Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland; Anja Lachenmayer, MD, Study Director — Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland; Vanessa Banz, MD PhD, Study Director — Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland; Daniel Candinas, Professor, MD, Study Chair — Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland
Locations (1):
- Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruix J, Reig M, Sherman M. Evidence-Based Diagnosis, Staging, and Treatment of Patients With Hepatocellular Carcinoma. Gastroenterology. 2016 Apr;150(4):835-53. doi: 10.1053/j.gastro.2015.12.041. Epub 2016 Jan 12. PMID 26795574
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Cho YK, Kim JK, Kim MY, Rhim H, Han JK. Systematic review of randomized trials for hepatocellular carcinoma treated with percutaneous ablation therapies. Hepatology. 2009 Feb;49(2):453-9. doi: 10.1002/hep.22648. PMID 19065676
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Bolondi L, Burroughs A, Dufour JF, Galle PR, Mazzaferro V, Piscaglia F, Raoul JL, Sangro B. Heterogeneity of patients with intermediate (BCLC B) Hepatocellular Carcinoma: proposal for a subclassification to facilitate treatment decisions. Semin Liver Dis. 2012 Nov;32(4):348-59. doi: 10.1055/s-0032-1329906. Epub 2013 Feb 8. PMID 23397536
- [Background] Wang X, Hu Y, Ren M, Lu X, Lu G, He S. Efficacy and Safety of Radiofrequency Ablation Combined with Transcatheter Arterial Chemoembolization for Hepatocellular Carcinomas Compared with Radiofrequency Ablation Alone: A Time-to-Event Meta-Analysis. Korean J Radiol. 2016 Jan-Feb;17(1):93-102. doi: 10.3348/kjr.2016.17.1.93. Epub 2016 Jan 6. PMID 26798221
- [Background] Lau WY, Lai EC. The current role of radiofrequency ablation in the management of hepatocellular carcinoma: a systematic review. Ann Surg. 2009 Jan;249(1):20-5. doi: 10.1097/SLA.0b013e31818eec29. PMID 19106671
- [Background] Sala M, Llovet JM, Vilana R, Bianchi L, Sole M, Ayuso C, Bru C, Bruix J; Barcelona Clinic Liver Cancer Group. Initial response to percutaneous ablation predicts survival in patients with hepatocellular carcinoma. Hepatology. 2004 Dec;40(6):1352-60. doi: 10.1002/hep.20465. PMID 15565564
- [Background] van Duijnhoven FH, Jansen MC, Junggeburt JM, van Hillegersberg R, Rijken AM, van Coevorden F, van der Sijp JR, van Gulik TM, Slooter GD, Klaase JM, Putter H, Tollenaar RA. Factors influencing the local failure rate of radiofrequency ablation of colorectal liver metastases. Ann Surg Oncol. 2006 May;13(5):651-8. doi: 10.1245/ASO.2006.08.014. Epub 2006 Mar 17. PMID 16538411
- [Background] Engstrand J, Toporek G, Harbut P, Jonas E, Nilsson H, Freedman J. Stereotactic CT-Guided Percutaneous Microwave Ablation of Liver Tumors With the Use of High-Frequency Jet Ventilation: An Accuracy and Procedural Safety Study. AJR Am J Roentgenol. 2017 Jan;208(1):193-200. doi: 10.2214/AJR.15.15803. Epub 2016 Oct 20. PMID 27762601
- [Background] Widmann G, Schullian P, Haidu M, Bale R. Stereotactic radiofrequency ablation (SRFA) of liver lesions: technique effectiveness, safety, and interoperator performance. Cardiovasc Intervent Radiol. 2012 Jun;35(3):570-80. doi: 10.1007/s00270-011-0200-4. Epub 2011 Jun 14. PMID 21671150
- [Background] Engstrand J, Nilsson H, Jansson A, Isaksson B, Freedman J, Lundell L, Jonas E. A multiple microwave ablation strategy in patients with initially unresectable colorectal cancer liver metastases - A safety and feasibility study of a new concept. Eur J Surg Oncol. 2014 Nov;40(11):1488-93. doi: 10.1016/j.ejso.2014.05.003. Epub 2014 May 20. PMID 24933395